CLINICAL TRIAL: NCT07311824
Title: Pain Management Optimization for In-Office Gynecologic Procedures: The Development and Evaluation of a Risk-Stratification Pain Calculator
Brief Title: Pain Management for In-Office Gynecologic Procedures Using a Risk-Stratification Pain Calculator
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carle Foundation Hospital (Other)
Responsible Party: Principal Investigator, Claire Aucoin, Co-Investigator, Carle Foundation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24CRU4052
Record Dates: First submitted 2025-12-02; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Pain Management; Patient Satisfaction; Gynecologic Procedures
Keywords: pain management; patient satisfaction; gynecologic procedures; IUD insertion; hysteroscopy; endometrial biopsy; colposcopy; ambulatory gynecologic procedures
MeSH Terms: conditions — Agnosia; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Calculator (Experimental): Participants will answer the Pain Calculator Questionnaire that will determine if they are low, moderate, or high risk for severe pain during their procedure. They will receive assigned pain medications based on their risk.
  Interventions: Other: Pain Calculator
- Control (No Intervention): Participants will have their pain management determined by the provider's best judgement, using shared decision making

INTERVENTIONS:
Other: Pain Calculator — The risk-stratification calculator, or the Pain Calculator, will be a questionnaire that the participant will answer with a research team member. The questions asked will include age, menopausal status, delivery history, history of certain gynecologic disorders, past experiences with gynecologic procedures, and anxiety about their upcoming procedure. Their answers will sort participants into low, moderate, and high risk groups. Each group will receive escalating pain medications for their procedure.
  Other Names: risk-stratification calculator; risk-stratification algorithm
  Arms: Pain Calculator

SUMMARY:
The goal of this clinical trial is to learn how using a risk-stratification calculator to determine the risk of a patient experiencing severe pain during an in-office gynecologic procedure and subsequently assigning pain medications to be used for the procedure based on risk, will affect patients' pain during these procedures. The main questions it aims to answer are:

* Does using pain medications determined by a risk-stratification calculator improve patients' pain scores during if-office gynecologic procedures?
* Does using pain medications determined by a risk-stratification calculator improve patient satisfaction?

Researchers will compare using the risk-stratification calculator to decide on pain medications to a provider using their best judgement to decide on pain medications. This will help determine if patients have improved pain scores and satisfaction if they have their pain medications assigned using the risk-stratification calculator.

Participants who are undergoing a relevant in-office gynecologic procedure will:

* Receive pain medications for their procedure either based on their answers to questions for the risk-stratification calculator or based on their provider's best judgement.
* Answer an online survey about their experience with the procedure and related pain management.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Proficient in English
* Access to personal smart devices (smartphone, tablet, laptop, etc.)
* Will be undergoing the following in-office gynecologic procedures: IUD insertion, endometrial biopsy, colposcopy with cervical biopsy, or hysteroscopy

Exclusion Criteria:

* Under the age of 18
* Non-English-Speaking
* Have contraindications to taking NSAIDs, acetaminophen, lidocaine or its derivatives, or opioids
* Patients who are taking methadone, Suboxone, and/or naltrexone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Average Perceived Pain Score | At time of procedure and at 10 minutes after procedure
  Participants will rank their pain perceived during their procedures from 0, equivalent to no pain, to 10, equivalent to worst imaginable pain.
Participant Satisfaction with Procedure | At time of procedure
  Participants will rank their satisfaction with their experience during the procedure using a standard Likert Scale, ranging from 1, not at all satisfied, to 5, highly satisfied.

SECONDARY OUTCOMES:
Average Perceived Pain Stratified by Risk Group | At time of procedure and at 10 minutes after procedure
  Using the same pain scale - 0 (no pain at all) to 10 (worst imaginable pain), pain scores of experimental group participants stratified by Risk Group will be each compared to the control group.
Participant Satisfaction with Procedure Stratified by Risk Group | at time of procedure
  Using the same Likert Scale - 1 (not at all satisfied) to 5 (highly satisfied), experimental group participants stratified by Risk Group will each be compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly London, MD, Principal Investigator — Carle Foundation Hospital; Georgina Cheng, MD PhD, Principal Investigator — Carle Foundation Hospital
Locations (2):
- United States (2):
  - Carle Champaign on Curtis, Champaign, Illinois
  - Carle Foundation Hospital, Urbana, Illinois

IPD SHARING:
Plan to Share IPD: No